CLINICAL TRIAL: NCT05841095
Title: Phase I/II Study to Determine the Safety, Immunogenicity and Efficacy of the Therapeutic Hepatitis B Virus Synthetic Long Peptide Vaccination ISA104
Brief Title: Evaluation of the Novel Therapeutic Hepatitis B Virus Synthetic Long Peptide Vaccination ISA104
Acronym: HEB-PEP
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Erasmus Medical Center (Other)
Collaborators: ISA Pharmaceuticals B.V. (Industry)
Responsible Party: Principal Investigator, Dave Sprengers, Priniciple Investigator, MD PhD, Erasmus Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MEC22-0600
Record Dates: First submitted 2023-03-27; First posted 2023-05-03 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Chronic Hepatitis b
Keywords: Immunotherapy; Therapeutic Vaccination; Hepatitis B cure
MeSH Terms: conditions — Hepatitis B, Chronic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ISA104 (Active Comparator)
  Interventions: Drug: ISA104
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ISA104 — SLP vaccine
  Arms: ISA104
Drug: Placebo — Saline solution (0.9% NaCl)
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to test ISA104 in patients with chronic hepatitis B. The main question[s] it aims to answer are:

* How safe is ISA104?
* Does ISA104 induce immunity against hepatitis B virus?

Different doses of the vaccine ISA104 will be administered to participants. These participants are chronic HBV patients being actively treated with antiviral drugs.

Researchers will compare the ISA104 vaccine to a placebo.

ELIGIBILITY:
Inclusion Criteria:

* cHBV
* Active treatment with NUCs and HBV DNA < limit of quantification

Exclusion Criteria:

* Immune-compromised
* Evidence of liver cirrhosis

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2023-08-04 (Actual); Primary Completion 2024-09-01 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
Safety according to AEs, SAEs | 6 months
  AEs, SAEs

SECONDARY OUTCOMES:
HBV specific Immunogenicity- following ISA104 vaccination | 6 months
  Number of IFN-y Elispots per well after 3 day stimulation with SLPs will correspond to immunogenicity. Elispots will be performed before (baseline) and after treatment
Efficacy of ISA104 vaccination by using conventional biomarkers | 6 monts
  Levels of HBsAg, HBsAb, HBeAg, HBV DNA

OTHER OUTCOMES:
To study novel HBV disease markers in the study patient population to assist with treatment decisions and/or therapy response monitoring in general | 6 months
  Levels of HBcrAg

CONTACTS AND LOCATIONS:
Overall Officials: Dave Sprengers, MD, PhD, Principal Investigator — Erasmus Medical Center
Locations (1):
- Erasmus MC, Rotterdam, Netherlands

IPD SHARING:
Plan to Share IPD: No